CLINICAL TRIAL: NCT01969188
Title: A Study of Novel Immune Modulating Biomarkers in Patients With Spondyloarthritis With Axial Involvement
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014-227
Record Dates: First submitted 2013-06-14; First posted 2013-10-25 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-01

CONDITIONS: Spondyloarthritis
Keywords: spondyloarthritis; ankylosing spondylitis; psoriatic arthritis
MeSH Terms: conditions — Spondylarthritis; Spondylitis, Ankylosing; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SpA in RA: Patients with SpA with psoriatic arthritis (PsA), ankylosing spondylitis (AS), no biologic therapy for 3 months, over 18 yrs old.

SUMMARY:
Spondyloarthritis refers to a set of inflammatory disorders that mainly afflict the spine, joints and ligaments. A subtype of spondyloarthritis is Ankylosing Spondylitis - now known as axial spondyloarthropathy - which is characterized by inflammation of the joints in the spinal column, and the part of the back where the spine meets the pelvis. Another subtype of spondyloarthritis is Psoriatic Arthritis where patients often develop raised patches of reddened skin. The disease can advance to one of more joints in the body resulting in pain, swelling and stiffness. These forms of inflammatory arthritis can become chronic and over time can lead to pain, disability and deformity.

There is now evidence that patients with inflammatory arthritis that are diagnosed and treated earlier in the course of their symptoms may have better results. Yet although we know that early treatment is important, the investigators still don't know if there are factors that can predict how an individual patient's disease will progress over time in terms of losing mobility. The investigators also do not know the relationship between loosing mobility and the formation of bone around the spine and joints.

The investigators are doing this study because the investigators want to learn more about patients with these forms of arthritis - Ankylosing Spondylitis and Psoriatic Arthritis. The investigators want to learn more about the factors that can predict how their disease might progress over time and what their response to treatment might be. The investigators would also like to determine the proportion of patients with these types of symptoms and describe the best treatment strategies for them.

DETAILED DESCRIPTION:
The condition to be studied is Spondyloarthritis (SpA). The investigators will gather a cohort of patients with variants of SpA (n = 70), including Ankylosing Spondylitis (AS) and Psoriatic Arthritis (PsA) who have axial disease and fully characterize disease activity. Care guidelines suggest that these patients are seen at least twice within the first year with annual visits thereafter. Radiographs are desirable to assess disease progression, but are not always required. Treatment options for both PsA and AS patients include non-steroidal anti-inflammatory drugs (NSAIDs), steroid injections, disease modifying anti rheumatic drugs (DMARDs) and biologics (i.e. tumor necrosis factor inhibitors aka TNF inhibitors or TNFi's). The cohort of patients eligible for enrollment in this study would be those patients who for the preceding 6 weeks have not received biologic treatment such as infliximab,and who for the preceding 4 weeks have not received biologic treatments such as adalimumab, etanercept,golimumab, certolizumab pegol and other biologic therapies.

Subjects will be evaluated 4 times over two years: at enrollment, 24 weeks, 52 weeks and 104 weeks (with a 12 week window around each visit). Usual care for patients with SpA would include regular assessments of pain, function and mobility, assessments of spine and joint motion, joint swelling and tenderness with treatment changes at each follow up visit to reduce pain, improve function, address adverse events to medications and enhance spinal mobility. Interventions might include physical therapy, analgesics, NSAIDs, DMARDs or biologic therapies. The investigator would not assign specific interventions to the subjects of the study. All of this would be recorded.

Specific clinical information will be gathered at each visit using validated indexes and data collection instruments, including disease activity [using the Bath AS Disease Activity Index (BASDAI) and Ankylosing Spondylitis Disease Activity Score (ASDAS)], function (using the Bath AS Functional Index (BASFI), measure joint/ligament involvement, measuring tender and swollen joint counts, dactylitis, enthesitis (as quantified using the Spondyloarthritis Research Consortium of Canada (SPARCC) enthesitis index and spine involvement (measured as range of movement in the spine and hips using the Bath AS Metrology Index (BASMI).

ELIGIBILITY:
Inclusion Criteria:

* Patients with SpA should have a BASDAI of > 3.5 with radiographic evidence and a BASDAI of > 4 without radiographic evidence
* No biologic therapy for ≥ 4-6 weeks. Patients may have had a TNFi > 6 weeks prior to study entry, but patients currently receiving, for example, adalimumab, etanercept, infliximab, golimumab, certolizumab pegol or who have taken any TNFis within the previous 4-6 weeks are ineligible. They must have been off of Remicade for 6 weeks, and off all other Biologics for 4 weeks.
* ≥18 yrs old
* Diagnosis of Spondyloarthritis (SpA) (per the Assessment of SpondyloArthritis(ASAS) criteria and having sacroiliitis as confirmed by radiographs or MRI at baseline), with psoriatic arthritis (PsA) (per the ASAS or Classification Criteria for Psoriatic Arthritis(CASPAR) criteria).
* Patients must have evidence of sacroiliitis either by radiograph or MRI, or must have evidence of spine inflammation confirmed by radiographs or spine MRI

Exclusion Criteria:

* Patients currently receiving biologic therapy (e.g. adalimumab, etanercept, infliximab, golimumab, certolizumab pegol)
* Diagnosis of a systemic rheumatic disease or crystalline arthritis (i.e. Rheumatoid Arthritis(RA), Systemic Lupus Erythematosus(SLE), systemic sclerosis, gout, pseudogout, Lyme arthritis, reactive arthritis, viral arthritis)
* Pregnant or nursing
* Unable to give informed consent
* Lack of fluency in English. Unfortunately, we do not have the financial resources to offer full translation services
* Unwilling or unable to be followed as part of routine care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of spondloarthritis with axial involvement and no biologic treatment in most recent three months (see inclusion criteria).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2013-01; Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Correlation between the change in IL-23R(Interleukin-23 receptor) levels and disease activity at one year and two years. | 12 months and 24 months.
  The primary outcome will be the correlation between IL-23R levels measured by flow cytometry with disease activity in patients with SpA as measured by the ASDAS, at one year and at two years.

SECONDARY OUTCOMES:
Difference in peripheral blood IL-23R levels in "responders", and correlation of other immune modulators and inflammatory cytokines | 12 months and 24 months
  (a) A secondary outcome will be the difference in peripheral blood IL-23R levels in patients whose ASDAS improves by at least 1.1 over 1 year and will be measured at the end of the first year and again at the end of the two-year study period. These patients will be referred to as "responders" to usual care. (We will also look at changes in level of IL-23R over 2 years in responders vs. non responders). A change of at least 1.1 is the minimally clinically important difference.
  b) We will evaluate the correlation of other immune modulators and inflammatory cytokines such as, TNF, IL-1, IL-6, IL-17, IL-22, and IL-21 and disease activity in patients who are followed serially with standard disease activity measures (ASDAS, BASDAI), function (BASFI), and enthesitis (MASES)(1, 2).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- See also: Hospital for Special Surgery — http://www.hss.edu
- See also: Principal Investigator, Vivian Bykerk MD — http://www.hss.edu/physicians_bykerk-vivian.asp